CLINICAL TRIAL: NCT06806891
Title: Restless Leg Syndrome: Is There a Response to Buddhist Walking Meditation in Hemodialysis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of physical therapy for Cardiovascular, Respiratory disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005557
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Hemolysis; Restless Legs Syndrome
MeSH Terms: conditions — Hemolysis; Restless Legs Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group number 1 (Experimental): the participants will be on hemodialyis. they complain restless leg syndrome. the participants will receive Buddhist walking meditation. this program of meditation will be 30 minutes thrice weekly. before and after Buddhist walking meditation .. the number of patients in the group will be 20. the total duration of Buddhist walking meditation will be 12 weeks.
  Interventions: Behavioral: Buddhist walking meditation
- group number 2 (No Intervention): the participants will be on hemodialyis. they complain restless leg syndrome. the number of patients in the group will be 20. this group will be control group that will not receive training .

INTERVENTIONS:
Behavioral: Buddhist walking meditation — the participants will be on hemodialyis. they complain restless leg syndrome. the participants will receive Buddhist walking meditation. this program of meditation will be 30 minutes thrice weekly. before and after Buddhist walking meditation .. The number of patients in the group will be 20. the total duration of Buddhist walking meditation will be 12 weeks.
  Arms: group number 1

SUMMARY:
the restless leg syndrome is a common complaint in person who undergo hemodialysis. Buddhist walking meditation efficacy was not investigated in those population

DETAILED DESCRIPTION:
the total participants will be 40. all patients will be on hemodialyis. they complain restless leg syndrome. the participants will be divided to group I which received Buddhist walking meditation. this program of meditation will be 30 minutes thrice weekly. before and after buddhist meditation walking, there will be 5 minutes stretching exercises working as warm up or cooling down respectively. the other group will serve as control one .. the number of patient in every group will be 20. the total duration of Buddhist walking meditation will be 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* hemodialysis patient (40)
* complain of restless leg syndrome
* non obese patients

Exclusion Criteria:

* cardiac patients
* chest diseases
* mental diseases
* hepatic diseases
* lower limb orthopedic hurting

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — self-representation of gender identity.
Enrollment: 40 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2025-03-06 (Estimated); Study Completion 2025-03-06 (Estimated)

PRIMARY OUTCOMES:
international RLS Study Group Rating | it will be measured after 12 weeks
  it will assess the severity of the problem (restless leg syndrome)

SECONDARY OUTCOMES:
Pittsburg sleep quality index | it will be measured after 12 weeks
  it will assess sleep quality
fatigue severity scale | it will be measured after 12 weeks
  it will assess fatigue level
sit to stand test | it will be measured after 12 weeks
  it will assess number of sit to stand in 30 seconds
physical component of short form 12 | it will be measured after 12 weeks
  a questionnaire will assess physical abilities of patients
mental component of short form 12 | it will be measured after 12 weeks
  a questionnaire will assess mental status of patients
beck depression inventory | It will be measured after 12 weeks
  a questionnaire will assess depression status of patients
Trait Anxiety Inventory | it will be measured after 12 weeks
  it will assess anxiety in patients
diatolic blood pressure | it will be measured after 12 weeks
  it will be assessed manually
systolic blood pressure | it will be measured after 12 weeks
  it will be assessed manually
cortisol | It will be measured after 12 weeks
  it will be measured in serum
C reactive protein | It will be measured after 12 weeks
  it will be measured in serum
nitric oxide | It will be measured after 12 weeks
  it will be measured in serum

CONTACTS AND LOCATIONS:
Overall Officials: Ali MA Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- faculty of physical therapy Cairo university, Dokki, Giza Governorate, Egypt